CLINICAL TRIAL: NCT02481479
Title: SCARF: Saxagliptin on CArdiac StRucture and Function
Brief Title: Saxagliptin and Cardiac Structure and Function
Acronym: SCARF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-267
Record Dates: First submitted 2015-06-16; First posted 2015-06-25 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group -Paired comparison (Other): Saxagliptin 2.5mg or 5mg od
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — Eligible patients will undergo baseline CMR, commence treatment and then after 6 months undergo repeat CMR
  Other Names: Onglyza
Drug: Saxagliptin — Eligible patients will undergo baseline echocardiogram, commence treatment and then after 6 months undergo repeat echocardiogram
  Other Names: Onglyza
Drug: saxagliptin — Eligible patients will undergo baseline venipuncture, commence treatment and then after 6 months undergo repeat venipuncture
  Other Names: Onglyza

SUMMARY:
Diabetes is associated with a substantially increased risk of heart failure, which is associated with substantial morbidity and mortality. Despite the development of new therapeutic strategies to improve glycemic control, recent clinical data from the saxagliptin assessment of vascular outcomes recorded in patients with diabetes mellitus-thrombolysis in myocardial infarction (SAVOR-TIMI) 53 study observed an unexpected finding of an excess of adjudicated heart failure hospitalizations. This excess occurred in the setting of pre-existing heart failure (HF) hospitalization and in those with elevated biomarkers for heart failure such as N terminal pro Brain type natriuretic peptide (NT-pro BNP). A wealth of preclinical data did not suggest a mechanistic basis for an excess of heart failure events, however these preclinical studies primarily focused upon prevention based strategies as opposed to regression studies once established heart failure was present. This proposal seeks to understand if and how dipeptidyl peptidase-4 inhibitors (DPP4i,specifically saxagliptin) may influence the development of heart failure, by evaluating changes in cardiac structure and function using cardiac magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
The cardiovascular safety and potential cardioprotective effects of diabetes drugs have been the focus of recent research. Currently, the Food and Drug Administration (FDA) requires all new anti-diabetic drugs to demonstrate no important increase in cardiovascular adverse events before approval.

Dipeptidyl peptidase-4 (DPP-4) inhibitors (gliptins) are oral incretin-based agents that increase glucagon-like peptide-1 (GLP-1) level, with proven anti-hyperglycemic effects and are increasingly used in the management of type 2 diabetes. In a rat model of diabetes and myocardial infarction, sitagliptin treatment improved passive left ventricular compliance, increased endothelial cell density, reduced myocyte hypertrophy and collagen abundance. GLP-1 and DDP-4 inhibition with vildagliptin improve cardiac function, cardiac remodeling, and survival in animal models of pressure-overload and chronic heart failure. However, in another study of post-MI cardiac remodeling in mice, vildagliptin failed to show any early or late protective effects on cardiac function.

Some clinical studies suggest that GLP-1 infusion is associated with an absolute increase in left ventricular ejection fraction (LVEF) in patients with heart failure, although data are conflicting. The GLP-1 receptor analog, exenatide may reduce infarct size in patients with myocardial infarction but does not improve LVEF.

The Cardiovascular Outcomes Study of Alogliptin in Patients With Type 2 Diabetes and Acute Coronary Syndrome EXAMINE trial randomized assigned 5340 patients with type 2 diabetes and recent acute coronary syndrome to alogliptin or placebo, and found no increase in adverse cardiovascular events in the alogliptin group. In SAVOR-TIMI 53, 16,492 patients with type 2 diabetes who had a history of, or were at risk for, cardiovascular events were randomized to receive saxagliptin or placebo. Over a median follow-up of 2.1 years, the primary composite endpoint of cardiovascular death, myocardial infarction, or ischemic stroke did not differ significantly between the 2 groups (P=0.99 for superiority; P<0.001 for noninferiority). However, patients in the saxagliptin group were more likely to be hospitalized for heart failure, which was not ascertained in the EXAMINE trial. Furthermore, the Sitagliptin Cardiovascular Outcome Study (TECOS), which examined the DPP4i sitagliptin versus placebo in high risk patients for a cardiovascular event demonstrated cardiovascular safety (P<0.001 for non inferiority), and there was no signal for excess heart failure hospitalizations.

Cardiac magnetic resonance imaging (CMR) has emerged as the "gold standard" for measuring LV volume, mass, and ejection fraction. LV volume measurements by cardiac MRI do not rely on geometric assumptions. CMR measurements have excellent intra-observer, inter-observer, and inter-study variability, which were superior to other imaging techniques. The high inter-study reproducibility of CMR affords a substantial reduction in the required sample size to demonstrate even small changes in LV volume, LV mass or LVEF, or conversely, to reliably exclude clinically important changes. Furthermore, CMR tagging allows detailed and quantitative assessment of regional LV diastolic and systolic function. For example, in the Multiethnic Study of Atherosclerosis (MESA), CMR can detect subtle alterations in global and regional LV functions in patients with traditional and novel cardiovascular risk factors. Although prior studies have failed to demonstrate any beneficial effects of improved glycemic control on myocardial function, CMR promises to be a more sensitive and accurate technique.

Accordingly, the investigators propose to use CMR to examine the cardiac structure, global and regional function among patients with type 2 diabetes treated with saxagliptin.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) men or women with type 2 diabetes diagnosed for ≥ 6 months
2. HbA1c 7.5 - 9.5%
3. Receiving background therapy with metformin (additional anti-hyperglycemic agents are permitted)
4. Clinical decision to initiate saxagliptin to improve glycemic control, as per treating physician

Exclusion Criteria:

1. GLP-1 receptor agonist or DPP4 inhibitor treatment within the past 6 months, or known intolerance
2. eGFR <30
3. Baseline LVEF <40%
4. NYHA Class III-IV or recent hospitalization for decompensated HF (<3 months)
5. Unstable coronary syndromes or recent revascularization within the past 3 months, or planned revascularization in the next 6 months
6. Significant (moderate or severe, or symptomatic) valvular disease
7. Pregnancy/childbearing potential
8. Routine contraindications to CMR Subjects who drop out from the study will have a repeat CMR examination as soon as possible after drug discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
The change in LVEF from baseline to 6 months | baseline, 6 months
  assess LVEF at baseline and at 6 months following treatment. CMR based LVEF assessment using Cvi 42.

SECONDARY OUTCOMES:
The change in E/e' from baseline to 6 months | baseline, 6 months
  Echocardiography assessed E and E', to determine ratio, and assess change from baseline to 6 months.
change in class indicators of signs and symptoms of heart failure at each visit | baseline, 6 months
  assess NYHA class at baseline and at 6 months
Change in log-scale in NT-pro BNP | baseline, 6 months
  assess NT-ProBNP at baseline and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, Study Director — Professor of Surgery
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 yr
Access Criteria: contact study PI